CLINICAL TRIAL: NCT00213148
Title: A Phase II, Prospective, Randomized, Double-Blind, Multicenter, Dose Finding, Comparative Study for the Evaluation of the Aromatase Inhibitor Anastrozole (Multiple-Dose) Versus Clomiphene Citrate in Stimulating Follicular Growth and Ovulation in Infertile Women With Ovulatory Dysfunction
Brief Title: Comparison of Anastrozole Verses Clomiphene Citrate in Stimulating Follicular Growth and Ovulation in Infertile Women With Ovulatory Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25550
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2017-09

CONDITIONS: Anovulation
MeSH Terms: conditions — Anovulation | interventions — Anastrozole; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Clomiphene Citrate 50 Milligram (mg) (Active Comparator)
  Interventions: Drug: Clomiphene Citrate 50 mg
- Clomiphene Citrate 100 mg (Active Comparator)
  Interventions: Drug: Clomiphene Citrate 100 mg
- Anastrozole 1 mg (Experimental)
  Interventions: Drug: Anastrozole 1 mg
- Anastrozole 5 mg (Experimental)
  Interventions: Drug: Anastrozole 5 mg
- Anastrozole 10 mg (Experimental)
  Interventions: Drug: Anastrozole 10 mg

INTERVENTIONS:
Drug: Anastrozole 1 mg — Subjects will be administered orally with 1 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month).
  Arms: Anastrozole 1 mg
Drug: Anastrozole 5 mg — Subjects will be administered orally with 5 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month).
  Arms: Anastrozole 5 mg
Drug: Anastrozole 10 mg — Subjects will be administered orally with 10 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month).
  Arms: Anastrozole 10 mg
Drug: Clomiphene Citrate 50 mg — Subjects will be administered orally with 50 mg of clomiphene citrate once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month).
  Arms: Clomiphene Citrate 50 Milligram (mg)
Drug: Clomiphene Citrate 100 mg — Subjects will be administered orally with 100 mg of clomiphene citrate once daily for 5 days in Cycle 2 and 3 (each cycle = approximately 1 month).
  Arms: Clomiphene Citrate 100 mg

SUMMARY:
The purpose of this study is to investigate and compare the safety and efficacy of various doses of the aromatase inhibitor (anastrozole) versus clomiphene citrate in stimulating follicular growth and ovulation in infertile women with ovulatory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years
* Ovulatory dysfunction characterized by irregular and/or extended cycles
* Non-smoker

Exclusion Criteria:

* No previous gonadotropin treatment
* No more than 6 previous clomiphene treatment cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2005-03-10 (Actual); Primary Completion 2007-12-12 (Actual); Study Completion 2007-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (1):
- Local US Medical Information, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clomiphene Citrate 50 Milligram (mg): Subjects were administered orally with 50 mg of clomiphene citrate once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month). Subjects in this arm were re-randomized at the start of Cycle 2 and Cycle 3 and either continued receiving Clomiphene Citrate 50 mg or moved to Clomiphene Citrate 100 mg arm.
- Clomiphene Citrate 100 mg: Subjects from Clomiphene Citrate 50 mg arm who were re-randomized at the start of Cycle 2 and Cycle 3 and were administered orally with 100 mg of clomiphene citrate once daily for 5 days in Cycle 2 and 3 (each cycle = approximately 1 month) were presented.
- Anastrozole 1 mg: Subjects were administered orally with 1 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month). Subjects in this arm were re-randomized at the start of Cycle 2 and Cycle 3 and either continued receiving Anastrozole 1 mg or moved to Anastrozole 10 mg arm.
- Anastrozole 5 mg: Subjects were administered orally with 5 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month). Subjects in this arm were re-randomized at the start of Cycle 2 and Cycle 3 and either continued receiving Anastrozole 5 mg or moved to Anastrozole 10 mg arm.
- Anastrozole 10 mg: Subjects were administered orally with 10 mg of anastrozole once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month). Some of the subjects from Anastrozole 1 mg and 5 mg arms were re-randomized at the start of Cycle 2 and Cycle 3 to Anastrozole 10 mg arm.
Period: Cycle 1 (1 Month)
Arm/Group | Clomiphene Citrate 50 Milligram (mg) | Clomiphene Citrate 100 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg
Started | 77 | 0 | 79 | 76 | 39
Completed | 53 | 0 | 60 | 58 | 17
Not Completed | 24 | 0 | 19 | 18 | 22
Not completed — Lost to Follow-up | 1 | 0 | 2 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 8 | 5 | 8
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0
Not completed — Other | 3 | 0 | 2 | 2 | 7
Not completed — Pregnancy Unrelated to Therapy | 0 | 0 | 0 | 1 | 0
Not completed — Non Resolving Cyst > 25mm | 0 | 0 | 0 | 0 | 1
Not completed — Discontinued Before Start of Cycle 2 | 15 | 0 | 5 | 8 | 5
Period: Cycle 2 (1 Month)
Arm/Group | Clomiphene Citrate 50 Milligram (mg) | Clomiphene Citrate 100 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg
Started | 43 | 10 | 42 | 52 | 41
Completed | 29 | 4 | 28 | 33 | 11
Not Completed | 14 | 6 | 14 | 19 | 30
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2 | 1
Not completed — Lack of Efficacy | 1 | 3 | 7 | 6 | 16
Not completed — Other | 2 | 1 | 2 | 8 | 7
Not completed — Pregnancy Unrelated to Therapy | 0 | 1 | 0 | 0 | 0
Not completed — Non Resolving Cyst > 25mm | 1 | 0 | 0 | 0 | 0
Not completed — Discontinued Before Start of Cycle 3 | 10 | 1 | 3 | 3 | 6
Period: Cycle 3 (1 Month)
Arm/Group | Clomiphene Citrate 50 Milligram (mg) | Clomiphene Citrate 100 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg
Started | 23 | 10 | 26 | 24 | 22
Completed | 23 | 8 | 25 | 23 | 21
Not Completed | 0 | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clomiphene Citrate 50 mg: Subjects were administered orally with 50 mg of clomiphene citrate once daily for 5 days in Cycle 1, 2 and 3 (each cycle = approximately 1 month). Subjects in this arm were re-randomized at the start of Cycle 2 and Cycle 3 and either continued receiving Clomiphene Citrate 50 mg or moved to Clomiphene Citrate 100 mg arm.
- Total: Total of all reporting groups
Arm/Group | Clomiphene Citrate 50 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg | Total
Number analyzed (Participants) | 77 | 79 | 76 | 39 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (3.9) | 28.8 (3.9) | 29.6 (3.9) | 29.3 (3.4) | 29.2 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 79 | 76 | 39 | 271
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ovulation Rate in Cycle 1
Description: Ovulation rate was defined as the percentage of subjects who ovulated (mid-luteal Progesteron [P4] level greater than or equal to [>=] 10 nanogram per milliliter [ng/mL] and/or pregnancy).
Time Frame: Up to 1 month
Population: All Treated population included all treated subjects who received at least one tablet of study drug (clomiphene citrate or anastrozole).
Measure: Number; unit: percentage of subjects
Groups:
- Clomiphene Citrate 50 mg: Subjects were administered orally with 50 mg of clomiphene citrate once daily for 5 days in Cycle 1.
- Anastrozole 1 mg: Subjects were administered orally with 1 mg of anastrozole once daily for 5 days in Cycle 1.
- Anastrozole 5 mg; Anastrozole 10 mg: Subjects were administered orally with 5 mg of anastrozole once daily for 5 days in Cycle 1.
Arm/Group | Clomiphene Citrate 50 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg
Number analyzed (Participants) | 77 | 79 | 76 | 39
percentage of subjects | 64.9 | 30.4 | 36.8 | 35.9

2. Secondary Outcome: Number of Subjects With Clinical Pregnancy in Cycle 1
Description: Clinical pregnancy was defined as the existence of at least one ultrasonographically confirmed gestational sac in the uterus with fetal heart activity.
Time Frame: Up to 1 month
Population: All Treated population included all treated subjects who received at least one tablet of study drug (CC or anastrozole).
Measure: Number; unit: subjects
Arm/Group | Clomiphene Citrate 50 mg | Anastrozole 1 mg | Anastrozole 5 mg | Anastrozole 10 mg
Number analyzed (Participants) | 77 | 79 | 76 | 39
subjects | 10 | 4 | 7 | 0

ADVERSE EVENTS:
Groups:
- Clomiphene Citrate 50 mg (Cycle 1): Subjects administered orally with 50 mg of clomiphene citrate once daily for 5 days in cycle 1 were presented.
- Anastrozole 1 mg (Cycle 1): Subjects administered orally with 1 mg of Anastrozole once daily for 5 days in cycle 1 were presented.
- Anastrozole 5 mg (Cycle 1): Subjects administered orally with 5 mg of Anastrozole once daily for 5 days in cycle 1 were presented.
- Anastrozole 10 mg (Cycle 1): Subjects administered orally with 10 mg of Anastrozole once daily for 5 days in cycle 1 were presented.
- Clomiphene Citrate 50 mg (Cycle 2): Subjects administered orally with 50 mg of clomiphene citrate once daily for 5 days in cycle 2 were presented.
- Clomiphene Citrate 100 mg (Cycle 2): Subjects administered orally with 100 mg of clomiphene citrate once daily for 5 days in cycle 2 were presented.
- Anastrozole 1 mg (Cycle 2): Subjects administered orally with 1 mg of Anastrozole once daily for 5 days in cycle 2 were presented.
- Anastrozole 5 mg (Cycle 2): Subjects administered orally with 5 mg of Anastrozole once daily for 5 days in cycle 2 were presented.
- Anastrozole 10 mg (Cycle 2): Subjects administered orally with 10 mg of Anastrozole once daily for 5 days in cycle 2 were presented.
- Clomiphene Citrate 50 mg (Cycle 3): Subjects administered orally with 50 mg of clomiphene citrate once daily for 5 days in cycle 3 were presented.
- Clomiphene Citrate 100 mg (Cycle 3): Subjects administered orally with 100 mg of clomiphene citrate once daily for 5 days in cycle 3 were presented.
- Anastrozole 1 mg (Cycle 3): Subjects administered orally with 1 mg of Anastrozole once daily for 5 days in cycle 3 were presented.
- Anastrozole 5 mg (Cycle 3): Subjects administered orally with 5 mg of Anastrozole once daily for 5 days in cycle 3 were presented.
- Anastrozole 10 mg (Cycle 3): Subjects were administered orally with 10 mg of Anastrozole once daily for 5 days in cycle 3 were presented.
Arm/Group | Clomiphene Citrate 50 mg (Cycle 1) | Anastrozole 1 mg (Cycle 1) | Anastrozole 5 mg (Cycle 1) | Anastrozole 10 mg (Cycle 1) | Clomiphene Citrate 50 mg (Cycle 2) | Clomiphene Citrate 100 mg (Cycle 2) | Anastrozole 1 mg (Cycle 2) | Anastrozole 5 mg (Cycle 2) | Anastrozole 10 mg (Cycle 2) | Clomiphene Citrate 50 mg (Cycle 3) | Clomiphene Citrate 100 mg (Cycle 3) | Anastrozole 1 mg (Cycle 3) | Anastrozole 5 mg (Cycle 3) | Anastrozole 10 mg (Cycle 3)
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/79 | 0/76 | 0/39 | 0/43 | 0/10 | 0/42 | 0/52 | 0/41 | 0/23 | 0/10 | 0/26 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 23/77 | 12/79 | 17/76 | 4/39 | 6/43 | 2/10 | 2/42 | 4/52 | 7/41 | 4/23 | 2/10 | 1/26 | 2/24 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clomiphene Citrate 50 mg (Cycle 1) (N=77) | Anastrozole 1 mg (Cycle 1) (N=79) | Anastrozole 5 mg (Cycle 1) (N=76) | Anastrozole 10 mg (Cycle 1) (N=39) | Clomiphene Citrate 50 mg (Cycle 2) (N=43) | Clomiphene Citrate 100 mg (Cycle 2) (N=10) | Anastrozole 1 mg (Cycle 2) (N=42) | Anastrozole 5 mg (Cycle 2) (N=52) | Anastrozole 10 mg (Cycle 2) (N=41) | Clomiphene Citrate 50 mg (Cycle 3) (N=23) | Clomiphene Citrate 100 mg (Cycle 3) (N=10) | Anastrozole 1 mg (Cycle 3) (N=26) | Anastrozole 5 mg (Cycle 3) (N=24) | Anastrozole 10 mg (Cycle 3) (N=22)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clomiphene Citrate 50 mg (Cycle 1) (N=77) | Anastrozole 1 mg (Cycle 1) (N=79) | Anastrozole 5 mg (Cycle 1) (N=76) | Anastrozole 10 mg (Cycle 1) (N=39) | Clomiphene Citrate 50 mg (Cycle 2) (N=43) | Clomiphene Citrate 100 mg (Cycle 2) (N=10) | Anastrozole 1 mg (Cycle 2) (N=42) | Anastrozole 5 mg (Cycle 2) (N=52) | Anastrozole 10 mg (Cycle 2) (N=41) | Clomiphene Citrate 50 mg (Cycle 3) (N=23) | Clomiphene Citrate 100 mg (Cycle 3) (N=10) | Anastrozole 1 mg (Cycle 3) (N=26) | Anastrozole 5 mg (Cycle 3) (N=24) | Anastrozole 10 mg (Cycle 3) (N=22)
Headache (Nervous system disorders) | 9 | 5 | 9 | 2 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 5 | 2 | 2 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 6 | 2 | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other